CLINICAL TRIAL: NCT00552682
Title: Pilot, Opened, Randomized Clinical Trial to Assess the Efficacy of Duloxetine in the Treatment of Fibromialgy in Patients With Infection by HIV 1+
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIBROHIV
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia; HIV-1 Infection
Keywords: HIV; fibromialgy; chronic fatigue syndrome; duloxetine; pain; treatment experienced; Fibromialgy in patients with HIV-1 infection
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Duloxetine 60 mg, 1 tablet/day
  Interventions: Drug: Duloxetine 60 mg, QD
- B (No Intervention): To continue with the antidepressive treatment if exist

INTERVENTIONS:
Drug: Duloxetine 60 mg, QD — Duloxetine 60 mg, 1 table/day, 1 year
  Other Names: Xeristar
  Arms: A

SUMMARY:
The purpose of this study is to compare duloxetine with conventional treatment of pain in HIV-1 infected patients.

DETAILED DESCRIPTION:
Among HIV-1-infected patients, diagnosis of fibromialgy has increased over the last years . Appropriate identification of firomialgy in these patients is challenging and sometimes can be more complicated than in HIV-negative population. Concomitant infectious processes and symptoms due to HIV infection itself need to be ruled out before establishing a formal diagnosis.

The treatment of this disease frequently includes muscular relaxants , pain-killers, anti-inflammatories and antidepressives despite no drug is formally indicated for this pathology.

Duloxetine approved indications include both treatment of major depressive disorders (MDD) and diabetic neuropathic pain. Recent studies in HIV negative patients show efficacy to control pain and depressive symptoms in patients with fibromialgy The main purpose of this pilot study is to assess the efficacy of duloxetine in HIV-1-infected patients with fibromialgy.

The main purpose of this pilot study is to assess the efficacy of duloxetine in HIV-1-infected patients with fibromialgy or chronic fatigue syndrome presenting with widespread pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old and more. Age +18 years old.
2. Documented HIV-1-infection.
3. Former diagnosis of fibromialgy.
4. History of good compliance with visit schedule and medication intake.
5. Patients voluntary signed the informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding females
2. Suspicion of intolerance to duloxetine.
3. History of any clinical condition that, in the Investigator's criteria, could potentially reoccur with the suggested change of therapy (sarcoma, lymphoma, etc).
4. Concomitant condition that could mimic fibromialgy (lupus, endocrine diseases, muscular diseases, multiple sclerosis)
5. or Acute illness within 15 days prior to the inclusion
6. Patients with major depressive disorder with psychotic symptoms, major depressive disorder melancholic type or bipolar disorder. Patients with other depressive disorders can be included (dysthymic disorder and depressive disorder NOS)
7. Anorexia or nervous bulimia
8. History or suspected drug or alcohol abuse.
9. Glaucoma
10. History of heart disease including cardiac arrhythmias
11. Severe obesity (body mass index > 45).
12. Concomitant medication with IMAOS, cimetidine or quinolonas
13. Patients with hepatic or renal serious failure (Creatinin clearance <30 ml/min)
14. Patients with Hypericum perforatum as a concomitant treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Variation in pain measured using the Brief Pain Inventory questionnaire in both branches of the study | Time frame: basal visit, weeks 4, 12, 24, 36 and 48

SECONDARY OUTCOMES:
Assess differences in Short-Form 36 Health Survey (SF-36) questionnaire scale score. | basal visit, weeks 12, 24 and 48
Assess differences in Beck Depression Inventory (BDI) questionnaire scale score. | basal visit, weeks 12, 24 and 48
Assess differences in Profile of Mood States - Forma A (POMS-A) questionnaire scale score. | basal visit, weeks 12, 24 and 48
Assess the percentage of patients that leave duloxetine due to intolerance or toxicity. | basal visit, weeks 4, 12, 24, 36 and 48
Assess, if possible, pharmacokinetic profile of duloxetine and determine interaction with antiretroviral drugs. | basal visit, weeks 4, 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Negredo Eugenia, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain